CLINICAL TRIAL: NCT00551551
Title: Urinary Postpartum Handicap Prevention: Pelvic Floor Exercises vs Control. Multicentric Randomized Trial
Brief Title: Prenatal Pelvic Floor Prevention (3PN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: CIC-EC Réunion (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3PN; AFSSAPS-2007-A00641-52
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Urinary Incontinence; Anal Incontinence; Genital Prolapse
Keywords: Pelvic floor; Kegel exercises; Quality of Life; Pelvic Pain
MeSH Terms: conditions — Urinary Incontinence; Encopresis; Pelvic Pain | interventions — Physical Therapists

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rééducation (Experimental): Standardized pelvic floor muscle training program with a physiotherapist in 8 sessions (20-30 minutes each) between 24 and 36 weeks of gestation AND Written instructions about personal (Kegel) pelvic floor exercises
  Interventions: Other: Pelvic floor muscle training with physiotherapist; Other: Written information about kegel exercises
- Control (Active Comparator): Written instructions about personal (Kegel) pelvic floor exercises
  Interventions: Other: Written information about kegel exercises

INTERVENTIONS:
Other: Pelvic floor muscle training with physiotherapist — 8 sessions of 20-30 minutes each between 24 and 36 weeks of gestation with a physiotherapist or midwife
  Other Names: pelvic floor exercises; Pelvic Floor Muscle Training; pelvic floor physiotherapy
  Arms: Rééducation
Other: Written information about kegel exercises — Information about pelvic floor disorders prevention with personal pelvic floor exercises
  Other Names: kegel exercises

SUMMARY:
Objective: Compare pelvic floor disorders (urinary incontinence, anal incontinence, genital prolapse, perineal pain, sexual troubles) 12 month after a first delivery between a group of women with prenatal pelvic floor exercises and a control group.

Hypothesis: Prenatal pelvic floor exercises reduce postpartum urinary incontinence.

DETAILED DESCRIPTION:
Justification:

Pelvic floor disorders lead to handicap and medical care consumption. Pregnancy and delivery are the main etiologies. Pelvic floor exercises are proposed for prevention and may reduce immediate postpartum incontinence but we do not know if this preventive effect persists at 1 year.

Principal criteria:

* Urinary incontinence score at 12 months post-partum (ICIQ-SF)

Secondary criteria:

* Urinary incontinence prevalence at pregnancy end, 2 and 12 months post-partum
* Other pelvic floor disorders at pregnancy end, 2 and 12 months post-partum: symptoms questionnaires, QOL questionnaire, Pad-test, POP-Q.
* Mode of delivery, length of active second phase, perineal tears, Apgar score.
* Number of postpartum pelvic floor session, number of medical consultations, Kegel exercises.

Progress:

* Inclusion between 20 and 28 weeks, initial assessment, randomization.
* 8 sessions of pelvic floor exercises with a physiotherapist between 24 and 36 weeks versus written information only.
* Assessment at pregnancy end, 2 and 12 (+/-1) month post-partum

Study length:

* For each women 18 months.
* For each center 30 months.

Number of subjects:

* To show a 1 point difference on ICIQ-SF score, we need 182 subjects (sd=2,4, a=0,05, β=0,20 bilateral test).
* Taking in account lost of follow-up (estimated 1/3) we are going to include 280 women.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous
* aged 18 years or more
* pregnant between 20 and 28 weeks
* French language reader

Exclusion Criteria:

* No medical insurance
* multiple or pathologic pregnancy
* Previous pelvic floor exercises with a physiotherapist less than 6 months before pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2007-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence score assessed with ICIQ-SF questionnaire | one year post partum

SECONDARY OUTCOMES:
Urinary incontinence prevalence | pregnancy end, 2 and 12 months post partum
Other pelvic floor symptoms (anal incontinence, pain, sexual troubles) | pregnancy end, 2 and 12 months post partum
Genital prolapse assessed by POP-Q | 2 months post-partum
Pelvic floor strength | 2 months post partum
Quality of life (Euroquol 5D, Contilife) | at delivery, 2 and 12 months post partum
pad-test | 2 months post partum
need to medical care | 12 months post partum

CONTACTS AND LOCATIONS:
Overall Officials: Xavier FRITEL, MD, PhD, Principal Investigator — CHR Réunion, CH Félix Guyon
Locations (5):
- France (5):
  - CHR Réunion, CH Félix-Guyon, Saint-Denis, Réunion
  - CHU Antoine-Béclère, Clamart
  - CHU Clermont, Clermont-Ferrand
  - CHU Caremeau, Nîmes
  - CH Poissy-Saint-Germain, Saint-Germain

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Fritel X, de Tayrac R, Bader G, Savary D, Gueye A, Deffieux X, Fernandez H, Richet C, Guilhot J, Fauconnier A. Preventing Urinary Incontinence With Supervised Prenatal Pelvic Floor Exercises: A Randomized Controlled Trial. Obstet Gynecol. 2015 Aug;126(2):370-377. doi: 10.1097/AOG.0000000000000972. PMID 26241428